CLINICAL TRIAL: NCT04071574
Title: Comparative Study on the Efficacy of Ovarian Stimulation Protocols on the Success Rate of ICSI in Women With Infertility Problems
Brief Title: Comparative Study on the Efficacy of Ovarian Stimulation Protocols on the Success Rate of ICSI in Female Infertility
Acronym: CS-EOSP-ICSI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Nehman Makdissy, Professor, Lebanese University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LU-MC-001/18
Record Dates: First submitted 2019-08-13; First posted 2019-08-28 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Female Infertility; Female Infertility Due to Ovulatory Disorder; Premature Ovarian Failure; Polycystic Ovary Syndrome; Female Infertility of Tubal Origin; Ectopic Pregnancy; Salpingitis; Female Infertility Due to Tubal Block; Female Infertility Due to Tubal Occlusion; Hydrosalpinx; Female Infertility - Cervical/Vaginal; Female Infertility Endocrine; Endometriosis; Fibroids; Congenital Uterine Anomaly; Infections Uterine; Female Infertility of Other Origin
Keywords: Infertility; Ovarian; Ovulation; IVF; ICSI; Gonadotropin
MeSH Terms: conditions — Infertility, Female; Primary Ovarian Insufficiency; Polycystic Ovary Syndrome; Pregnancy, Ectopic; Salpingitis; Endometriosis; Leiomyoma; Uterine Anomalies; Endometritis; Infertility | interventions — Chorionic Gonadotropin; Gonadotropins; Menotropins; Triptorelin Pamoate; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; cetrorelix

STUDY DESIGN:
Intervention Model Description: comparative protocols
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Protocol "A" (Active Comparator): Protocol with gonadotropins alone without agonist or antagonist:
  Gonadotropin treatment begins after spontaneous menses. The gonadotropins (e.g. Menopur, 150-225IU) are injected daily from D2/3 of the cycle (Gonadotropin dose varies based on the follicular response). The moment to trigger ovulation by administration of HCG (e.g. Ovitrelle or Pregnyl, 10.000IU) is determined by monitoring ovulation (folliculogenesis) approximately 14 days after gonadotropins regimen and the presence of at least 3 follicles with 18 mm sizes and at least the levels of E2 reaches 250-300 pg/ml. 36 h after HCG triggering, the mature oocytes are retrieved.
  Interventions: Drug: Human Chorionic Gonadotropin (hCG); Drug: Gonadotropins
- Protocol "B" (Active Comparator): Short GnRH agonist protocol:
  For the short GnRH agonist protocol, the administration of gonadotropins begins at the same time as that of the agonist, which makes it possible to take advantage of the action of endogenous gonadotropins released by the flare-up effect of the agonist. A low dose of GnRH agonist (e.g., triptorelin (Decapeptyl 0.1mg/day)) is administered in parallel to gonadotropin (e.g. Menopur, 150-225 IU) daily starting on cycle-day 2 (Gonadotropin dose varies based on the follicular development). Continual administration of GnRH agonist and gonadotropin lasts until HCG triggering (e.g. Ovitrelle or Pregnyl, 10.000IU), ~14 days post GnRH agonist regimen when follicles size reached 16-18 mm and at least the levels of E2 reaches 250-300 pg/ml. 36 h after HCG triggering, the mature oocytes are retrieved.
  Interventions: Drug: Human Chorionic Gonadotropin (hCG); Drug: Gonadotropins; Drug: GNRH-A Triptorelin
- Protocol "C" (Active Comparator): Multiple-dose antagonist protocol:
  For the GnRH antagonist protocol, a low dose of GnRH antagonist (0.25 mg/day) is administered. The protocol starts with the administration of gonadotropin (e.g. Menopur, 150-225 IU) daily which is initiated after monitoring of patients' follicles sizes on cycle-day 2/3 (Gonadotropin dose varies based on the follicular response). Almost after the 6th days of gonadotropin injection or when follicular size reaches more than or equal to 14 mm, GnRH antagonist (e.g., cetrorelix (cetrotide) or ganirelix (orgulatron) 0.25mg) begins by subcutaneous administration every day till HCG triggering (e.g. Ovitrelle or Pregnyl, 10.000IU). 36 h after HCG triggering, the mature oocytes are retrieved.
  Interventions: Drug: Human Chorionic Gonadotropin (hCG); Drug: Gonadotropins; Drug: GnRH antagonist
- Protocol "D" (Active Comparator): Long GnRH agonist protocol:
  For the long GnRH agonist protocol, a low dose of GnRH agonist (e.g., triptorelin (Decapeptyl 0.1mg)) is administered on cycle-day 21 followed by gonadotropin (e.g. Menopur, 150-225 IU) daily starting on cycle-day 2 after menses (Gonadotropin dose varies based on the follicular development). Continual administration of GnRH agonist and gonadotropin lasts until HCG triggering (e.g. Ovitrelle or Pregnyl, 10.000IU), ~14 days post GnRH agonist regimen when follicles size reached 16-18 mm. 36 h after HCG triggering, the mature oocytes are retrieved.
  Interventions: Drug: Human Chorionic Gonadotropin (hCG); Drug: Gonadotropins; Drug: GNRH-A Triptorelin
- Protocol "E" (Active Comparator): Combined GnRH antagonist and agonist protocol:
  For the combined protocol, it starts with the administration of gonadotropin (e.g. Menopur, 150-225 IU) daily which is initiated after monitoring of patients' follicles sizes on cycle-day 2/3 (Gonadotropin dose varies based on the follicular response). Almost after the 6th days of gonadotropin injection or when follicular size reaches more than or equal to 14 mm, GnRH antagonist (e.g., cetrorelix (cetrotide) or ganirelix (orgulatron) 0.25mg) begins by subcutaneous administration every day till GnRH agonist injection (e.g., triptorelin (Decapeptyl 0.1mg/day)). 36 h after agonist injection, the mature oocytes are retrieved.
  Interventions: Drug: Gonadotropins; Drug: GNRH-A Triptorelin; Drug: GnRH antagonist

INTERVENTIONS:
Drug: Human Chorionic Gonadotropin (hCG) — Administration of hCG (10.000IU) for ovulation triggering
  Other Names: OVITRELLE / PREGNYL
  Arms: Protocol "A"; Protocol "B"; Protocol "C"; Protocol "D"
Drug: Gonadotropins — Administration of Menotropin (hMG / FSH and LH at a 1:1 ratio) (150-225IU/day)
  Other Names: MENOPUR
Drug: GNRH-A Triptorelin — Administration of Triptorelin (0.1mg/day)
  Other Names: DECAPEPTYL
  Arms: Protocol "B"; Protocol "D"; Protocol "E"
Drug: GnRH antagonist — Administration of cetrorelix (cetrotide) or ganirelix (orgulatron) (0.25mg/day)
  Other Names: CETROTIDE / ORGULATRON
  Arms: Protocol "C"; Protocol "E"

SUMMARY:
The study will describe the effectiveness of ovarian stimulation in correlation with female infertility causes in a Lebanese population: a comparative study using 5 protocols of ovulation induction (treatment with "A" gonadotropins alone, "B" short GnRH agonist, "C" multiple-dose GnRH antagonist, "D" long GnRH agonist and "E" combined protocol of GnRH antagonist and agonist) and the outcomes of ICSI. This comparative study will help clinicians to select the relevant protocol of ovarian stimulation related to the female infertility disorders.

DETAILED DESCRIPTION:
One in six couples worldwide is affected by infertility, which defined as the inability to conceive after one year or more of regular and unprotected intercourse. It has been stated that 48.5 million couples in the world, with unprotected coitus, suffer from infertility. In about 50% of them, the infertility is due to female factors and diseases associated with the female reproductive system. Epidemiological studies show that 10 to 15% of all married couples are estimated to have infertility problems in the Middle East. Lebanon, in particular, is characterized with traditional and westernized lifestyles; It has high rates of smoking and caffeine intake, pollution and high rates of consanguinity marriage (11 to 17%), which affect considerably the conception rate.

The desire to procreate is naturally present in women all over the world. Due to various advances in medical procreation techniques, it has become possible for many women to realize their hope. Women were more likely to be psychologically distressed to infertility and suffer from poor quality of life more than men once they are diagnosed as infertile.

The causes of female infertility can have a genetic, anatomical or physiological origin. Among the most common genetic causes of female infertility are the chromosomes abnormalities: the numbers of X chromosomes, homogeneous or mosaic; other abnormalities are reciprocal translocations, Robertsonian translocations, inversions, supernumerary markers or abnormalities of the X chromosome structure. In such cases, no treatment and procreation require an egg donation. But the main causes of female infertility are physiological and anatomical, such as ovulatory disorders (25%), endometriosis (15%), pelvic adhesions (12%), tubal blockage (11%), other tubal abnormalities (11%), hyperprolactinemia (7%) and some minor causes. In addition, leiomyomas, fibroma, polyps, and tubal disease, may reduce fertility. In addition came the environmental factors (drugs, pesticides, food, tobacco ...) and there is an increase in the percentage of infertile women with advancing female age. A French national survey on lifestyles and toxic factors in infertile couples showed that in women, tobacco generates a risk twice as high as being infertile, a decrease in the ovarian reserve where the level of anti-Mullerian hormone (AMH) decreases, irregular short cycles and dysmenorrhea are also found in smokers. In addition, products contained in tobacco such as cotinine, cadmium and hydrogen peroxide are found in the follicular fluid and would be responsible for an alteration of the recovery of oocyte meiosis.

Couples who have problems with conception are referred to a medically assisted procreation (MAP) for fertility treatments. These treatments can be very stressful both psychologically and physically. Indeed, the numerous medical appointments and examinations, as well as the many bereavements and failures, experienced following repeated attempts at conception can to consume the married, social and professional life of couples. In addition, fertility issues require significant financial resources to cover the costs of fertility treatments, but also those related to the maternal and fetal complications of pregnancy, which are more frequent in the case of MAP pregnancies than in spontaneous conception.

Control of the ovarian stimulation is the key component of assisted reproductive technologies (ART) that have shifted the clinical practice of natural mono-follicular cycles into multi-follicular stimulated cycles. The increase in the number of follicles, and consequently the number of oocytes recovered, improved pregnancy rates in women undergoing In Vitro Fertilization (IVF) / Intra-Cytoplasmic Sperm Injection (ICSI), not only by increasing the number of available embryos but also by allowing embryo culture extended and allowing the selection of higher quality embryos to be transferred. However, several studies have addressed the issue of the optimal number of oocytes recovered following controlled ovarian stimulation (COS) for IVF / ICSI and demonstrated that the ovarian response is independently related to Live Birth Rate (LBR) after IVF / ICSI.

Many new treatment modalities for ovarian stimulation have been introduced over the years - often with insufficient evidence of safety and efficacy - using different compounds and regimens for ovarian stimulation, triggering oocyte maturation, interventions preceding stimulation supplementation phase. The most important clinical challenge is to find the right balance between improving the chances of success (birth of a healthy child), a reasonable cost, acceptable discomfort for the patient, and a minimal complication rate. New developments make ovarian stimulation less intense and more individualized. The choice of the ovarian stimulation protocol is one of the most important steps in IVF/ICSI treatment.

This study aims to identify and evaluate ovarian stimulation protocols applied to different patients with different causes of female infertility prior to medically assisted procreation techniques in order to know if there is a relationship between a given protocol and the result obtained for each class of infertility. Therefore, 360 ICSI in 200-300 couples will be studied in order to evaluate the link between ovarian stimulation protocols and outcomes of ICSI.

The population will be divided into 3 groups:

1. Group "OD" for ovulation disorders caused by endocrine disorders such as the polycystic ovarian syndrome (PCOS) and/or premature ovarian failure (POF)
2. Group "TD" for tubal disorders caused by previous ectopic pregnancy, salpingectomy, tubal obstruction and/or hydrosalpinx
3. Group "UCD" for uterine and cervical disorders caused by fibroids, endometriosis, infection and/or congenital uterine anomaly (CUA)

ELIGIBILITY:
Inclusion Criteria:

* must not show any of the excluded criteria
* Patients affected by female infertility due to particularly Ovulatory Disorder, Premature Ovarian Failure, Polycystic Ovary Syndrome, Tubal Origin, Ectopic Pregnancy, Salpingitis, Tubal Block/Occlusion, Hydrosalpinx, Cervical/Vaginal, Endocrine, Endometriosis, Fibroids, Congenital Uterine Anomaly, Infections Uterine, and Female Infertility of Other Origin
* The selection of subjects' age must be group matched between protocols of treatment. Premature ovarian failure is defined as AMH (Anti Mullerian Hormone) ≤ 2 ng/mL.
* Willing to collaborate and to attend to the clinical follow-ups for the next three years
* Patients willing to sign informed consent
* Able and willing to comply with all study requirements
* Absence of genetic causes
* Medically suitable to undergo ovarian stimulation
* Normal serum chemistry and hematology screening tests
* Negative human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV) serology
* No history of malignancy
* Complete history & physical examination

Exclusion Criteria:

* Subjects to be excluded from the study if the male (husband) had any male infertility problem(s)
* Patients with any genetic abnormalities
* Patients with histories of neurologic conditions including moderate or severe head injury, stroke, cerebral or bone damage or malignancies, brain abnormalities, learning disability, major medical or psychiatric illness, and metabolic/cardiovascular disease or evidence of cardiac/renal damage or malignancies, alcohol, loss of weight during the last 2 years, chemotherapy or immunosuppressive therapy.
* Women aged 45 years and older, under 21 years

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The average age of the population must be around 30 years old. Note that no one of the 264 women in this study should have any chromosomal abnormalities or mutated genes that affect ovarian function.
Enrollment: 200 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Ovulation Induction | 36 hours
  Monitoring of Ovulation Stimulation by trans-vaginal ultrasound determining the growth, number and appearance of the ovarian follicles as well as the maturation of the endometrium (measurement of its thickness); Follicles are considered mature when their diameter is greater than 18-20mm and each of them provides 250-300pg/mL of E2. When these criteria are obtained, ovulation is triggered

SECONDARY OUTCOMES:
fertilization rate | 12 months
  Changes in the fertilization rate
embryo quality | 12 months
  Selection of embryos for transfer depending on their morphology, and the regularity of blastomers
pregnancy rate | 12 months
  Determination of βHCG for positive results
live birth rate | 12 months
  Calculations of live birth rate are based on the number of live births in each group divided by all live births, multiplied by 100

CONTACTS AND LOCATIONS:
Overall Officials: Nehman Makdissy, Professor, Study Chair — Lebanese University; Samar El Hamoui, Dr, Study Director — Lebanese University
Locations (1):
- Lebanese University, faculty of sciences III, Tripoli, North Lebanon, Lebanon

IPD SHARING:
Plan to Share IPD: No